CLINICAL TRIAL: NCT02977338
Title: Evaluation in Patients With Obstructive Sleep Apnea That Had Undergone Diagnosis and Surgical Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0052-16-HYMC
Record Dates: First submitted 2016-11-10; First posted 2016-11-30 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-12

CONDITIONS: OSA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Retrospective review

SUMMARY:
Drug induced sleep endoscopy (DISE) is an increasingly performed procedure, offering dynamic upper airway evaluation during artificial sleep before surgical treatment for patients with obstructed sleep apnea (OSA).

DISE is a safe procedure, easily practicable, valid and reliable. The investigators consider it a fundamental clinical procedure that is essential before choosing the surgical treatment. The investigator's results so far suggest that a multilevel collapse is significantly associated with higher apnea hypopnea index values. The investigators think that the weight did not play a significant role in RDI reduction. Results till now show that tailored surgery based on DISE may leverage sleep surgeries outcome significantly, presenting 70% success rate based on the investigator's experience The aim of this study is to evaluate surgery results in patients who underwent DISE prior to their surgery in comparison to their condition prior to the treatment.

DETAILED DESCRIPTION:
Drug induced sleep endoscopy (DISE) is an increasingly performed procedure, offering dynamic upper airway evaluation during artificial sleep before surgical treatment for patients with obstructed sleep apnea (OSA).

Aim: To evaluate the value of DISE for tailoring the proper treatment for patients with snoring and OSA.

DISE is a safe procedure, easily practicable, valid and reliable. It is considered a fundamental clinical procedure that is essential before choosing the surgical treatment. Results so far suggest that a multilevel collapse is significantly associated with higher apnea hypopnea index values. The investigators think that the weight did not play a significant role in RDI reduction. Results till now show that tailored surgery based on DISE may leverage sleep surgeries outcome significantly, presenting 70% success rate based on the investigator's experience The aim of this tudy is to evaluate surgery results in patients who underwent DISE prior to their surgery in comparison to their condition prior to the treatment.

The results of the DISE based treatment will be compared with literature data from patients who underwent the surgery without DISE.

Method:

A retrospective follow-up study. Patients with snoring and OSA, had sleep study and had DISE before deciding on the surgical treatment. DISE findings were reported using the NOHL and VOTE classifications systems; site, degree of airway narrowing and configuration of obstruction. Patients underwent tailored surgery based on DISE findings included multi-level surgery; palate, tonsils, base of tongue and epiglottis.

After examining the results of the surgery in the patients, a comparison will be made based on sleep laboratory parameters (RDI, minimum saturation, degree of sleep apnea, degree of snoring) with data from the literature for patients who did not undergo DISE. On the whole, the degree of improvement in the patient's condition will be assessed.

We would like to show preference in surgery outcome in patients who were diagnosed using DISE.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Female or Male
* Fully diagnosed patients with OSA (including sleep laboratory) who are candidates for surgery as a treatment for their condition.

Exclusion Criteria:

* Patients who are not candidates for surgery as a treatment for their OSA.
* Patients with high surgical risk.
* Patients with hematological and oncological background.
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with snoring and OSA.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory Disturbance Index (RDI) | 12 months
minimum saturation | 12 month
degree of sleep apnea | 12 month
degree of snoring | 12 month

IPD SHARING:
Plan to Share IPD: Undecided